CLINICAL TRIAL: NCT01175915
Title: A Clinical Trial To Evaluate Reduning Injection in the Treatment of Mild Type of Hand, Foot, and Mouth Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Collaborators: Beijing University of Chinese Medicine (Other)
Responsible Party: Wei Xiao, Jiangsu Kanion Pharmaceutical Co.,Ltd
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200907001-3-1
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2010-08

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Mild type of hand, foot and mouth disease; Reduning Injection; Effectiveness; Safety
MeSH Terms: conditions — Hand, Foot and Mouth Disease; Mouth Diseases | interventions — reduning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Western therapy (Active Comparator)
  Interventions: Other: Western therapy
- Reduning Injection (Experimental)
  Interventions: Other: Reduning Injection
- Reduning Injection plus western therapy (Experimental)
  Interventions: Other: Reduning Injection plus western therapy

INTERVENTIONS:
Other: Western therapy — 1. Adopting physical cooling therapy, including physical cooling paste or warm bathing, when patient's body temperature is lower than 38.5 degree Celsius;
  2. Using Ibuprofen suspension when patient's temperature higher than 38.5 degree Celsius lasting for more than 2 hours;
  3. No specific treatment for tetter and ulcer, but Bingpeng powder, Watermelon tablet or frost for oral herpes.
  Intervention time: 3-7 days; Follow-up time: 3 days.
  Arms: Western therapy
Other: Reduning Injection — 1. Lifestyle counseling, vitamin supplementation if necessary, and non-use of antibiotics;
  2. Reduning Injection, 0.5~15ml, depending on patient's condition, IV per day, or according to the instruction;
  3. Using Ibuprofen suspension when patient's temperature higher than 39 degree Celsius lasting for more than 2 hours.
  Intervention time: 3-7 days; Follow-up time: 3 days.
  Arms: Reduning Injection
Other: Reduning Injection plus western therapy — 1. General treatment including lifestyle counseling, vitamin supplementation if necessary, non-use of antibiotics, and symptomatic treatment as follows;
  2. Symptomatic treatment by western therapy adopting the same plan in western therapy comparator group;
  3. Symptomatic treatment by Reduning Injection adopting the same plan in Reduning Injection experimental group.
  Intervention time: 3-7 days; Follow-up time: 3 days.
  Arms: Reduning Injection plus western therapy

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of Reduning Injection for mild type of hand-foot-mouth disease.

DETAILED DESCRIPTION:
By adopting a multi-center, prospective, randomized and controlled clinical trial, this study is aimed to evaluate the efficacy and safety of Reduning Injection in the treatment of mild type of Hand, Foot and Mouth Disease (HFMD), and to provide medical evidence of Reduning Injection for HFMD, especially to offer suggestions in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe hand-foot-mouth disease patients according to Hand-Foot-Mouth Disease Treatment Guidelines 2010 issued by China's Ministry of Health; More than 1/3 patients should be diagnosed by etiological examination.
* Less than 48 hours of occurrence of mild symptoms, with an armpit temperature of more than 37.5 degrees Celsius.
* Less than 48 hours of occurrence of tetter or herpes.
* Age of 1-13 years.
* Patients or their guardians agree to participate in this study and signed the informed consent form.

Exclusion Criteria:

* Complicated with other serious primary diseases in organ such as congenital heart disease, chronic hepatitis, nephritis and blood diseases, etc.
* With history of allergies on the experimental medicine, or severe allergies to other medicines.
* Using other western medicine or Chinese medicine for treating HFMD when consulted.
* Attending other clinical studies on HFMD after diagnosed.

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
time of bringing down the fever | 10 days
  Refering to the length of time to bring down the fever by 0.5 degrees Celsius after the medicine is taken.
time of body temperature going back to normal | 10 days
  Refering to the time of the armpit temperature of lower than 37.0 degrees Celsius, lasting for at least 24 hours, after the medicine is taken.

SECONDARY OUTCOMES:
time of symptom disappearance | 10 days
  Refering to the length of time when clinical symptoms and signs totally disappere after the medicine is used.
time of tetter disappearance | 10 days
  Refering to the length of time when the tetter due to HFMD disappears, characterised by scab(s) or dropping; and time of oral ulcer concrescence, etc.
dose and usage of medicine | 10 days
  Refering to the dose and frequency of using the medicine.
case severity rate | 10 days
  Refering to the ratio of patient with mild type of HFMD to severe type.
adverse reaction incidence | 10 days
  Calculated by adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xiao, Principal Investigator — Jiangsu Kanion Pharmaceutical Co., Ltd
Locations (6):
- China (6):
  - An'Hui Provincial Children's Hospital, Hefei, An'Hui
  - Fujian Provincial Quanzhou City Children's Hospital, Quanzhou, Fujian
  - The Fifth Hospital of Shijiazhuang City, Shijiazhuang, Hebei
  - Kaifeng Municipal Children's Hospital, Kaifeng, Henan
  - Hunan Provincial Children's Hospital, Changsha, Hunan
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality